CLINICAL TRIAL: NCT06153927
Title: Diagnostic Performance of On-site Automatic Coronary Computed Tomography Angiography-derived Fractional Flow Reserve
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: Keimyung University Dongsan Medical Center (Other); Inje University Ilsan Paik Hospital (Other); Chosun University Hospital (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Other Study IDs: D-2207-023-1337
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
Keywords: Computed Tomography-based Fractional Flow Reserve; Coronary Computed Tomography Angiography; Fractional Flow Reserve; Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with CCTA and FFR assessment: Patients with CAD who underwent CCTA, invasive coronary angiography, and FFR measurement will be included in this study.
  Interventions: Diagnostic Test: CT-FFR

INTERVENTIONS:
Diagnostic Test: CT-FFR — CT-FFR was calculated using HeartMedi+ 1.0 according to the manufacturer's instructions

SUMMARY:
The current study evaluated the diagnostic performance for myocardial ischemia of on-site automatic CCTA-derived FFR (CT-FFR) using a commercially available workstation as compared with invasive FFR as a reference. The diagnostic performance of CT-FFR was compared to that of CCTA diameter stenosis.

DETAILED DESCRIPTION:
This is a retrospective, multicenter, comparative, investigator-initiated study to evaluate the diagnostic performance of CT-FFR from routinely acquired CCTA data using the software HeartMedi+ 1.0 (AI Medic, Korea) to detect hemodynamically significant CAD. Patients who underwent CCTA within 90 days before invasive coronary angiography and FFR measurement will be screened in each participating center. After that, invasive coronary angiography, FFR data, and CCTA data will be anonymized and transferred to the independent core laboratories and analyzed in a blind fashion.

The presence of ischemia was defined as FFR ≤0.80. Anatomical obstructive stenosis was defined as diameter stenosis on CCTA ≥50%, and the diagnostic performance of CT-FFR and CCTA stenosis for ischemia was compared.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 20 years or older
* individuals who had undergone ≥ 64 multidetector row CCTA within 90 days before invasive coronary angiography and FFR measurement
* individuals who had not experienced any clinical events or significant clinical changes between the time of CCTA and invasive coronary angiography

Exclusion Criteria:

* previous coronary intervention or coronary bypass surgery in the target vessel
* invasive coronary angiography under unstable conditions
* previous myocardial infarction at target vessel territory
* congenital heart disease
* moderate or severe valvular heart disease
* previous valvular heart surgery
* left ventricular ejection fraction ≤40% or left ventricular hypertrophy
* previous cardiac device implantation
* body mass index >35 kg/m2
* poor FFR tracing quality
* no information on the position of the FFR pressure wire
* heart rate ≥100 beats/min during CCTA
* CCTA calcium score ≥1000
* no nitroglycerin prior to CCTA
* CCTA slice thickness >1.0 mm
* significant artifacts in CCTA

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CAD patients who underwent CCTA, invasive coronary angiography, and FFR measurement will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 332 (Actual)
Dates: Start 2022-05-26 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of CT-FFR | At the time of test
  Diagnostic accuracy of CT-FFR to detect hemodynamically significant CAD evaluated with an invasive FFR

SECONDARY OUTCOMES:
Spearman's correlation coefficient of CT-FFR with FFR | At the time of test
  Spearman's correlation coefficient of CT-FFR with FFR
Agreement between CT-FFR and FFR | At the time of test
  Bland-Altman analysis was used to demonstrate the agreement between CT-FFR and FFR.
Comparison of diagnostic performance of CT-FFR to that of CCTA stenosis | At the time of test
  Diagnostic performance to predict hemodynamically significant CAD included diagnostic accuracy, sensitivity, specificity, positive predictive value, and negative predictive value.
  A comparison of diagnostic performance was performed using McNemar's test or weight generalized score statistic as appropriate.
Comparison of discriminant ability of CT-FFR to that of CCTA stenosis | At the time of test
  Discriminant ability to predict hemodynamically significant CAD was assessed by the area under the receiver-operating characteristic curve (AUC).
  The AUCs were compared by Delong's test

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea